CLINICAL TRIAL: NCT03997266
Title: NICU Antibiotics and Outcomes Trial
Acronym: NANO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Michael Morowitz (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Michael Morowitz, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY20110298; R01HD097578 (NIH)
Record Dates: First submitted 2019-06-02; First posted 2019-06-25 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Microbial Colonization; Extreme Prematurity; Early-Onset Neonatal Sepsis; Late-Onset Neonatal Sepsis; Necrotizing Enterocolitis of Newborn; Death; Neonatal
Keywords: premature birth; human microbiome; antibiotics
MeSH Terms: conditions — Communicable Diseases; Neonatal Sepsis; Perinatal Death; Premature Birth | interventions — Ampicillin; Gentamicins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empiric antibiotics (Active Comparator): Infants will receive standard antibiotic coverage of ampicillin and gentamycin at site approved dosing guidelines while completing an evaluation for early-onset neonatal sepsis.
  Interventions: Drug: Ampicillin; Drug: Gentamycin
- Placebo (Placebo Comparator): Infants will receive a volume matched placebo of normal saline while completing an evaluation for early-onset neonatal sepsis.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ampicillin — Intravenous ampicillin
  Arms: Empiric antibiotics
Drug: Gentamycin — Intravenous gentamycin
  Arms: Empiric antibiotics
Drug: Normal saline — Intravenous normal saline
  Arms: Placebo

SUMMARY:
The goal of the NANO trial is to study the longstanding clinical practice of empirically administering intravenous antibiotics to extremely low birthweight (ELBW) infants in the first days of life. In this 802-subject multicenter placebo-controlled randomized clinical trial, the hypothesis to be tested is that the incidence of adverse outcomes is higher in babies receiving empiric antibiotics (EA) in the first week of life compared to babies receiving placebo. The study targets a population of ELBW infants in whom the clinical decision to use or not use EA is currently most challenging -- infants that are clinically stable that did not have a known exposure to intraamniotic infection and were not born preterm for maternal indications. The primary outcome is the composite outcome of late-onset sepsis (LOS), necrotizing enterocolitis (NEC), or death during the index hospitalization. Secondary safety outcomes will include total antibiotic days, days to full enteral feedings, and common morbidities in preterm infants that have previously been linked to EA, e.g. retinopathy of prematurity and bronchopulmonary dysplasia. Weight and length z-score, and head circumference, are standard measures to be collected weekly by clinical team per a standardized protocol.

DETAILED DESCRIPTION:
Randomization and blinding. Physicians will screen infants based on inclusion/exclusion criteria. The site coordinator will confirm eligibility with the treating physician and input patient data into the web based system. Once data is inputted, the coordinator will randomize eligible families 1:1 using web-based block randomization stratified by study site to receive EA or placebo. Multiples (i.e. siblings) will be randomized to the same treatment arm. Randomization will be sent to the investigational pharmacy via email, where study drug will be drawn. Participants, treating clinicians, and study staff will all be blinded to allocation. Outcome assessors and statistical summaries for trial monitoring will be unaware of group allocation. Unblinded data evaluation during the trial will be restricted to a designated study statistician and the Data and Safety Monitoring Board (DSMB). Investigators will be unblinded and analyses initiated only after all data collection forms are completed, data queries resolved, and data are locked for analysis.

Intervention. Following randomization, the coordinator will contact the attending physician, nurse practitioner and/or other providers as appropriate, and nurse to inform them that randomization has been completed. The intervention consists of administering either conventional EA or placebo while completing an evaluation for early onset sepsis. Timing of drug administration will be closely monitored. Enrolled subjects will receive EITHER ampicillin and gentamicin at site approved dosing guidelines OR volume matched equivalent of normal saline. These dosing regimens are derived from updated published guidelines for neonates. No masking is required as each of these solutions is clear.

The study drug will be ordered and in many cases discontinued just as EA would normally be ordered and discontinued; specifically, this means that the drugs will be ordered and administered within 4 hours of life and then discontinued at the discretion of the attending neonatologist. Typically this occurs when blood culture results are deemed negative (expected in > 95% of study subjects). The study protocol will allow the first dose of study drug to be administered as late as 4 hours after delivery. Research coordinators will follow daily orders on all study subjects.

Fecal sample collection. Samples will be obtained exclusively for research purposes, and there will be no testing of patients beyond obtaining microbiome samples, and recording demographic data and clinical history. Spontaneously expelled fecal samples for microbiome analyses will be obtained weekly from study subjects through the first 8 weeks of life, and monthly thereafter until death or discharge.

Infant blood draw. An additional research blood sample for genetic analysis will be drawn one time and should be done at the time of clinical blood draws. However, if this blood draw is missed, it can be done in the neonate's first week of life. A volume of 0.3 to 0.4mL will be drawn in EDTA tubes and shaken well. After the sample is collected, it will be frozen for shipment. The blood draw will be performed by NICU personnel who routinely draw blood on preterm babies. It will be either the bedside nurse or the respiratory therapist depending on whether the blood is drawn from an umbilical catheter or by heelstick.

Maternal vaginal swab and rectal swabs at delivery will be collected. If a rectal swab was not collected at the time of delivery, a maternal fecal sample during the first week postpartum will be collected in its place. Samples will be cryopreserved at -80C.

An electronic database will be used to track sample collection and storage history.

ELIGIBILITY:
I. Inclusion criteria: We will enroll newborn infants with gestational age of 23-30 weeks 6 days infants at participating study sites will be eligible.

II. Exclusion criteria:

1. Infants born for maternal indications via caesarean section with rupture of membranes at delivery, without attempts to induce labor, and without concern for maternal infection
2. Infants at high risk of EOS

   * Infants born to mothers with intrapartum fever (> 38C) or clinical diagnosis of chorioamnionitis
   * Infants born to mothers with previous infant with GBS disease/infection
3. Infants with respiratory insufficiency requiring invasive mechanical ventilation and FiO2 > 0.40 or non-invasive ventilation and FiO2 > 0.60 at time of randomization
4. Infants with ongoing hemodynamic instability requiring vasopressors or fluid boluses at time of randomization
5. Clinician concern infant is at high risk for sepsis due to infant physical exam findings or clinical history of mother or infant
6. Major congenital anomalies
7. Infants not anticipated to survive beyond 72 hours
8. Infants who have received antibiotics prior to randomization
9. Mothers that are <18 years old at time of enrollment

Max Age: 4 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 802 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Composite incidence of NEC, LOS, or death | From the time and day of randomization through the subject's date of death from any cause or discharge from the birth hospital, whichever comes first, assessed up until 50 weeks.
  NEC will be assessed by clinical presentation and an abdominal x-ray obtained and read by a certified radiologist. NEC will be defined strictly by Bell's stage II or III criteria for moderate or advanced NEC. To reduce overlap between NEC and diagnosis of spontaneous intestinal perforation, the diagnosis of NEC will only be considered in infants > 7 days of age. LOS is defined as defined as a positive blood culture obtained after 72 hours of life and intent to treat with antibiotics for 5 days or more. Death is defined as death during the index hospitalization.

SECONDARY OUTCOMES:
NEC | From the time and day of randomization through the subject's date of death from any cause or discharge from the birth hospital, whichever comes first, assessed up until 50 weeks.
  NEC will be assessed by clinical presentation and an abdominal x-ray obtained and read by a certified radiologist. NEC will be defined strictly by Bell's stage II or III criteria for moderate or advanced NEC. To reduce overlap between NEC and diagnosis of spontaneous intestinal perforation, the diagnosis of NEC will only be considered in infants > 7 days of age.
LOS | From the time and day of randomization through the subject's date of death from any cause or discharge from the birth hospital, whichever comes first, assessed up until 50 weeks.
  LOS is defined as defined as a positive blood culture obtained after 72 hours of life and intent to treat with antibiotics for 5 days or more.
Death | From the time and day of randomization through the subject's date of death from any cause or discharge from the birth hospital, whichever comes first, assessed up until 50 weeks.
  Death is defined as death during the index hospitalization.

OTHER OUTCOMES:
Microbial diversity within infant fecal samples | Weekly stool samples will be collected for the first 8 weeks of life and then monthly through death or discharge from the subject's birth hospital , assessed up to 50 weeks.
  Bacterial DNA will be sequenced according to established protocols. In analyses of these samples, we shall investigate three important parameters, namely, alpha diversity (Richness and Shannon Index), beta diversity, and the differential abundance of individual bacterial taxa.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - USA Children's and Women's Hospital, Mobile, Alabama
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of South Flordia Health, Tampa, Florida
  - University of Louisville Research Foundation Inc./Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - The Trustees of Columbia University in the City of New York, New York, New York
  - Golisano Children's Hospital at University of Rochester, Rochester, New York
  - Maria Fareri Children's Hospital at Westchester Medical Center, Valhalla, New York
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Penn State Medical College, Hershey, Pennsylvania
  - Pennsylvania Hospital/The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Alfred I. duPont for Children of the Nemours Foundation, Philadelphia, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morowitz MJ, Katheria AC, Polin RA, Pace E, Huang DT, Chang CH, Yabes JG. The NICU Antibiotics and Outcomes (NANO) trial: a randomized multicenter clinical trial assessing empiric antibiotics and clinical outcomes in newborn preterm infants. Trials. 2022 May 23;23(1):428. doi: 10.1186/s13063-022-06352-3. PMID 35606829